CLINICAL TRIAL: NCT02963948
Title: A Phased-Implementation Feasibility and Proof-of-Concept Study to Assess Incorporating the NIDA CTN Common Data Elements (CDEs) Into the Electronic Health Record (EHR) in Large Primary Care Settings ("CDE-EHR-PC" Study), Phase 3
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Massachusetts General Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-01373; CTN-0062Ot (Other: NIDA)
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Clinic A1
  Interventions: Behavioral: Meetings with implementation leader(s); Behavioral: the SAAS survey; Behavioral: Patient surveys
- Clinic A2
  Interventions: Behavioral: Meetings with implementation leader(s); Behavioral: the SAAS survey; Behavioral: Patient surveys
- Clinic B1
  Interventions: Behavioral: Meetings with implementation leader(s); Behavioral: the SAAS survey; Behavioral: Patient surveys
- Clinic B2
  Interventions: Behavioral: Meetings with implementation leader(s); Behavioral: the SAAS survey; Behavioral: Patient surveys
- Clinic B3
  Interventions: Behavioral: Meetings with implementation leader(s); Behavioral: the SAAS survey; Behavioral: Patient surveys
- Clinic B4
  Interventions: Behavioral: Meetings with implementation leader(s); Behavioral: the SAAS survey; Behavioral: Patient surveys

INTERVENTIONS:
Behavioral: Meetings with implementation leader(s) — The perceived appropriateness of the intervention to medical staff will affect an intervention's initial adoption as well as sustainability. We will assess this through focus groups with staff, conducted approximately 1-2 months after implementation of the screening and CDS tools.
Behavioral: the SAAS survey — Medical staff will be surveyed using the Substance Abuse Attitude Survey (SAAS) to gather information about attitudes from medical staff who do not participate in the focus groups, or may be uncomfortable sharing negative attitudes in a group of their peers. The SAAS is a validated multidimensional instrument that evaluates physician attitudes toward substance-using patients. It includes specific measures of attitudes toward permissiveness, treatment intervention, stereotypes, treatment optimism, and moralism, and has been used in prior studies of primary care physicians. Collecting information on staff attitudes toward substance users and substance use interventions will be helpful to inform about any sources for low adoption of the tools, and any needs for additional provider education and training.
Behavioral: Patient surveys — Patient surveys regarding attitudes toward substance use screening and interventions in the primary care clinic will be distributed to patients presenting for care, regardless of whether they completed screening, at regular time periods throughout this study phase. The survey will be conducted for 1 week at the following approximate intervals following successful implementation: 1 month, 4 months, 7 months, and 10 months

SUMMARY:
This is a 4-phase study to implement the NIDA CDEs in primary care settings. Collecting and utilizing the CDEs in clinical practice requires a strategy for implementing screening to collect substance use information that populates the CDEs, and assisting primary care medical staff to offer appropriate interventions by providing clinical decision support (CDS) and a mechanism for making referrals to addiction treatment. Investigators aim to maximize the efficient adoption of screening, CDS, and treatment referrals by integrating all of these activities into the electronic health record (EHR).

The study will be conducted at three sites, representing three large health systems. Each phase will include deliverables essential to move to the next phase, and an independent Advisory Committee will review progress and make recommendations at each transition about how best to progress to each subsequent phase. Based on progress during earlier phases, the Advisory Committee may recommend expansion to additional clinics or health systems during the second part of Phase 4.

DETAILED DESCRIPTION:
SPECIFIC AIMS

1. To program the NIDA CTN CDEs, the NIDA/ASAM electronic Clinical Quality Measure (eCQM), and a lean decision support module into Epic.
2. To study the process of implementation of screening and referral using Epic-driven CDEs and CDS in three primary care clinics / practices, including defining potential barriers and facilitators to their adoption.
3. To evaluate the impact of implementation on:

   * Patient level outcomes (diagnosis, treatment referral);
   * Medical staff level outcomes (screening and assessment, clinical interventions including counseling and treatment referral); and
   * Systems level outcomes (logistics and costs of introducing the CDEs, feasibility).

ELIGIBILITY:
Inclusion Criteria:

* English speaking adult individuals age 18 years or older, and current employee or patient at a Wave 1 clinic with direct patient contact.

Exclusion Criteria:

* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Number of subjects:
  * Approximately 40 medical staff will be enrolled for the focus groups
  * Approximately 100 medical staff will be surveyed using Substance Abuse Attitude Survey (SAAS)
  * Approximately 200 patients at a Wave 1 clinic
  Clinical implementation leaders Clinical implementation leaders are practicing primary care physicians (PCPs) who provide feedback to the research team and support their colleagues on implementing screening, using the CDS, and carrying out clinical interventions and referrals to address unhealthy substance use. One or two primary care providers will be identified from each participating clinic will advise the research team on implementation and to serve as a resource for their colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 113123 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Adoption of screening | 12 Months
  % patients presenting for primary care visits who were screened in the past 12 months
Provider adoption of CDS | 12 Months
  % patients with positive screens for which CDS was launched and completed
Referral of high risk patients | 12 Months
  % patients with high risk use who received referral to specialty care

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, PhD, Principal Investigator — New York University Medical School
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Result] McNeely J, Adam A, Rotrosen J, Wakeman SE, Wilens TE, Kannry J, Rosenthal RN, Wahle A, Pitts S, Farkas S, Rosa C, Peccoralo L, Waite E, Vega A, Kent J, Craven CK, Kaminski TA, Firmin E, Isenberg B, Harris M, Kushniruk A, Hamilton L. Comparison of Methods for Alcohol and Drug Screening in Primary Care Clinics. JAMA Netw Open. 2021 May 3;4(5):e2110721. doi: 10.1001/jamanetworkopen.2021.10721. PMID 34014326